CLINICAL TRIAL: NCT02733575
Title: A Case Series Study of Compassion Focused Therapy for Distressing Experiences
Brief Title: Compassion Focused Therapy for Distressing Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R&D2018/024
Record Dates: First submitted 2016-02-25; First posted 2016-04-11 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compassion Focused Therapy (Other): Intervention
  Interventions: Other: Compassion Focused Therapy

INTERVENTIONS:
Other: Compassion Focused Therapy — Up to 26 sessions of Compassion Focused Therapy

SUMMARY:
This study aims to develop and test the feasibility of a new therapy called Compassion Focused Therapy (CFT) for psychosis. This therapy helps people with psychosis manage distressing experiences by building internal feelings of safeness and affiliation, and by providing contexts, practices and insights that facilitate the development of compassion to self and others. The focus is on helping people feel safe in relation to their experiences and their social worlds. CFT is a promising new approach that has been successfully provided for people with a range of mental health difficulties. It is also firmly based in the most up-to-date knowledge and science about how the mind works (both normally and under stress).

9 participants will be recruited from NHS psychological therapies services for people with psychosis in South London and Maudsley (SLAM) NHS Foundation Trust. Following a short baseline period they will receive up to 26 weekly sessions (about 6 months) of CFT with a clinical psychologist, and will provide interview and questionnaire research data at five different points during the study. At these assessment points, data will be gathered on participants' experiences, mood, perceptions of their position in the social world, and heart rate variability.

The initial therapy protocol has been developed by psychologists with expertise in CFT, alongside people with lived experience of hearing voices and having distressing beliefs. However, it will continue to be developed and evolve as the study progresses, and as more is learnt (e.g. from the service-user participants) about applying the model in this population. At the end of this study, the aim is to have all the information needed to run a randomised controlled trial of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Psychosis related diagnosis (F20-39)
* Distressing positive symptoms of psychosis. Each participant will have been routinely screened with PSYRATS at their service entry assessment. On PSYRATS, at least one positive symptom (i.e. hallucination or delusion) will be present, and distress will be evidenced by an associated intensity score of 2 or above
* Willing to engage in psychological therapy
* Sufficient command of English language
* Able to provide informed consent

Exclusion Criteria:

* Currently engaged in CBT, or have completed a 12+ session course of CBT within the last 3 years. If recruitment is under target, this will be relaxed to 12+ session course of CBT (Cognitive Behavioural Therapy) within the last 6 months
* Currently engaged with another treatment study (e.g. medicine or therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Attrition rate measured by number dropping out of therapy | 6 months

SECONDARY OUTCOMES:
Psychotic symptoms measured by PSYRATS | Over 6 months of therapy, and 6-8 weeks post-therapy
  Measured by PSYRATS (Psychotic Symptom Rating Scales)
Depression and anxiety symptoms measured by DASS-21 | Over 6 months of therapy, and 6-8 weeks post-therapy
  Measured by DASS-21 (Depression, Anxiety and Stress Scale)
Subjective wellbeing, symptoms, functioning, and risk/harm measured by CORE | Over 6 months of therapy, and 6-8 weeks post-therapy
  Measured by CORE (Clinical Outcomes in Routine Evaluation)
Dissociative experiences measured by DES-II | Over 6 months of therapy, and 6-8 weeks post-therapy
  Measured by DES-II (Dissociative Experiences Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Heriot-Maitland, DClinPsych, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom